CLINICAL TRIAL: NCT00225316
Title: Can Maternal Acupuncture for Chemically Dependent Pregnant Women Reduce the Severity of Neonatal Abstinence Syndrome? - A Randomized Controlled Trial
Brief Title: Maternal Acupuncture for Substance Abuse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Patricia Janssen, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W05-0041; 04-2985
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Substance Addiction
Keywords: RCT; intervention study; addiction; substance use; pregnancy
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Acupuncture — See Detailed Description.

SUMMARY:
To determine the efficacy of daily maternal acupuncture treatments in reducing the frequency and severity of neonatal abstinence syndrome among infants born to substance-using women..

DETAILED DESCRIPTION:
Potential study subjects will be recruited from the Chemical Dependency Unit by a trial coordinator. After obtaining written informed consent, the coordinator will take a sequentially numbered opaque envelope from a box on the unit. This envelope will contain a card indicating the treatment group to which the woman is allocated. Women participating in the treatment group of our study will have access to a quiet room furnished with comfortable reclining chairs. The acupuncturist will swab the ears with alcohol and insert sterile, disposable needles. Following the treatment, which is 45-minutes in length, participants will remove the needles themselves and place them in protective sharps boxes. A sham acupuncture procedure will not be used. Chinese traditional medicine does not include the concept of a placebo. Those who argue that auricular acupuncture stimulates the vagus nerve, which innervates the ear concha state that needles placed anywhere in the concha should produce the same effects. 58 Studies utilizing sham procedures have failed to show a difference between the control and active experimental conditions.

In this unit, morphine is prescribed for the neonate by pediatricians (11 in total) if there is a constellation of symptoms unresponsive to environmental control including: 1) convulsions, 2) inconsolability or crying continuously for 3 hours, 3) persistent tremors or jitteriness when undisturbed, 4) continuous central nervous system irritability including hyperactive Moro reflex, tremors, jitteriness, increased muscle tone and unprovoked muscle jerks, 5) persistent vomiting or projectile vomiting over a 12 hour period; or 6) explosive diarrhea for 2-3 consecutive episodes. Additional clinical signs such as tachycardia, tachypnea, watery stools, fever, or weight loss > 10% may justify use of morphine after consideration of differential diagnoses. Morphine 1mg/ml is started at a rate of 0.03 mg/kg/dose every 3 hours. The dose is reviewed daily and titrated based on daily weights and ongoing symptoms.

ELIGIBILITY:
Inclusion Criteria:

Women admitted to the chemical dependency unit at BC Women's Hospital, Vancouver, B.C.

Exclusion Criteria:

* Women who neither read nor write English
* Having a pacemaker or any other electrical implants
* Bleeding disorder or on anti-coagulants
* Conditions putting someone at particular risk for infection including damaged heart valves or prior heart valve surgery, history of myocardiopathy, diabetes requiring insulin, history of knee or hip replacements, immunosuppressive drug therapy, open wounds.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Days of newborn morphine treatment

SECONDARY OUTCOMES:
Gestational age at birth, rates of intrauterine growth restriction, days to regain birthweight, rates of admission to a level II or level III nursery and length of stay, and rates of apprehension of the infant by the Ministry of Children and Families

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Patricia Janssen, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada